CLINICAL TRIAL: NCT06270303
Title: The Use of a Bone Substitute Material in the Surgical Therapy of Furcation Defects - a Multi-center Randomized Controlled Trial
Brief Title: Use of a Bone Substitute Material in the Surgical Therapy of Furcation Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other); Charite University, Berlin, Germany (Other); King's College London (Other); Queen Mary University of London (Other); Geistlich Pharma AG (Industry); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-00383-01
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis; Furcation Defects
Keywords: Surgical therapy; Reconstructive; Randomized controlled trial
MeSH Terms: conditions — Periodontitis; Furcation Defects

STUDY DESIGN:
Intervention Model Description: The project will be conducted as a two-armed randomized controlled trial in multiple clinical centers. The primary outcome will be assessed at 1 year post-surgery with a subsequent follow-up of 10 years.
Who Masked: Outcomes Assessor
Masking Description: Clinical assessments following intervention will be conducted by assessors unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Access flap + bone substitute (Experimental): Furcation defect will be treated by access flap debridement followed by application of a bone substitute material.
  Interventions: Procedure: Access flap & surgical debridement; Procedure: Application of bone substitute material (BioOss Collagen)
- Access flap (Active Comparator): Furcation defect will be treated by access flap debridement alone.
  Interventions: Procedure: Access flap & surgical debridement

INTERVENTIONS:
Procedure: Access flap & surgical debridement — Following surgical exposure, roots are carefully debrided.
Procedure: Application of bone substitute material (BioOss Collagen) — Following surgical debridement, the bone substitute material is applied to the furcation defect.
  Arms: Access flap + bone substitute

SUMMARY:
The aim of this randomized clinical trial is to evaluate the potential benefit of the use of a bone substitute material in the treatment of furcation degree II-involved molars. The main question it aims to answer is: What is the benefit of the adjunctive use of a bone substitute material in the surgical treatment of furcation degree II-involved molars when compared to open-flap debridement alone?

200 patients with ≥1 molar presenting with a furcation defect degree II will be included and randomized to either control (open-flap debridement) or test treatment (open-flap debridement + bone substitute material). The primary outcome of the study is furcation closure defined as absence of clinically detectable furcation involvement degree >I. Secondary outcomes include changes in bleeding on probing, probing depth, vertical and horizontal attachment levels, soft tissue level, marginal bone level, need for surgical retreatment, tooth loss, patient-reported outcomes and adverse events. A composite outcome based on furcation closure (degree ≤I) in combination with shallow probing depth (≤5 mm) and absence of bleeding on probing will also be evaluated.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled trial with a 12-month follow-up at multiple clinical centers throughout Europe. All study-related procedures are to be performed by specialists in periodontics or clinicians in specialist training. 200 patients with ≥1 molar with a furcation defect degree II (pre-surgical assessment) will be enrolled in the study. Following the primary evaluation at 12 months, study participants will be followed up to 10 years.

Preparatory phase Prior to surgery, patients will be provided with tailored non-surgical periodontal therapy including instructions in self-performed plaque control measures and supra- and subgingival instrumentation. The preparatory phase is concluded by an examination 8-16 weeks after completion of the non-surgical instrumentation.

Surgical intervention Following local anesthesia, full thickness flaps at target molars will be elevated and inflamed tissues are removed. Root surfaces are then instrumented using an ultra-sonic device with a standardized tip under irrigation with saline. Upon completion of root instrumentation, group allocation is revealed and a bone substitute material will be placed in the furcation defect to the level of the outer contour of the roots in the test group. Flaps will be repositioned and sutured to cover the entirety of the furcation area aiming for primary closure. The same procedure, omitting the placement of the bone substitute material, will be performed in the control group.

Patients will refrain from mechanical self-performed plaque control measures in the surgical area for 4 weeks post-surgery. During this period, daily rinsing with a 0.2% solution of chlorhexidine digluconate is prescribed.

Follow-up Sutures will be removed after two weeks and patient-reported experience (PRE) is scored. Patients will then be seen for oral hygiene instructions at 4 weeks and for supportive periodontal therapy at 3, 6, 9 and 12 months. Treatment and patient-reported outcomes (PROs) will be evaluated at 6 and 12 months. Additional examinations are carried out at 3, 5, 7 and 10 years.

Clinical assessments Clinical examinations at baseline and during follow-up will be performed by calibrated and blinded examiners. The following parameters will be recorded at all included teeth: degree of furcation, horizontal and vertical attachment levels. Bleeding on probing and plaque (yes/no), and probing pocket depth (mm), will be scored. Soft tissue levels will be assessed relative to the cemento-enamel junction.

During the surgical intervention, dimensions of the furcation defect will be noted. Adverse events will be noted

Radiographic assessments Standard intra-oral radiographs will be obtained at baseline, at 12 months and at years 3, 5 and 10. Assessments with regard to bone level changes and interradicular bone fill will be performed by an examiner blinded to group allocation.

Biomarkers In a nested approach, two centers (Gothenburg & London) will perform evaluations of inflammatory markers during healing. Prior to the surgical intervention and at 2 weeks, 6 months and 12 months, samples of gingival crevicular fluid (GCF) will be obtained. GCF will be collected at the target site as well as the contra-lateral molar (or alternative tooth if missing) utilizing PerioPaper strips. Inflammatory markers (eg IL-1, IL-6) will be evaluated through ELISA.

Questionnaire Patients will be asked to complete an assisted questionnaire at baseline, as well as at 6 and 12 months (PROs). Questions addressing patient satisfaction and potential discomfort after treatment are answered by means of a visual analogue scale (10 cm). Patient-reported experiences (PREs) will be scored at the 2-week control visit following the surgical intervention.

Enrolment, randomization, group allocation and blinding Patients meeting the inclusion criteria following completion of the preparatory phase will be invited on a consecutive basis. Upon signed consent, participants are enrolled and assigned a unique identification number, by which patients are randomly allocated to one of two study arms. Randomization (ratio 1:1) is performed by computer-generated lists with permuted blocks of eight and stratified for smoking. Allocation is concealed by the use of opaque envelopes not opened until completion of the surgical debridement. Examiners at baseline and during follow-up will be blinded to group allocation.

Data analysis Categorical and continuous variables originating from the clinical, radiographic and biomarker assessments will be evaluated by regression analyses adjusted for group allocation, time point (repeated measurements: baseline, 6 months, 1 year, etc.), smoking and tooth/furcation location (site; 1st vs 2nd molar; mandible vs maxilla). An intention-to-treat approach will be followed. It is assumed that drop-out will occur at random. Hence, latest available data points will be moved forward. A potential center effect will be evaluated. PROs are expected to be not-normally distributed and will be assessed through non-parametric methods.

ELIGIBILITY:
Inclusion Criteria:

Patients should present with at least one surgically accessible molar (in tooth position 6 or 7) diagnosed with a single furcation defect degree II (at any aspect).

Following initial periodontal therapy, teeth to be included should present with one site with furcation defect degree II in combination with:

* Bleeding on probing
* Probing pocket depth of ≥6 mm
* Soft tissue coverage of the furcation entrance Patients should present with a full mouth plaque score ≤25%.

Exclusion Criteria:

* Multiple deep furcation defects (degree II - III) at the same tooth
* Vertical attachment loss >50% at aspects not facing the furcation defect
* Defects presenting with apico-marginal communication
* Intake of systemic antibiotics within 6 months
* Systemic conditions/medication impeding surgical intervention (e.g. uncontrolled diabetes, immunosuppressive medication)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients/teeth displaying furcation closure. | 6 months.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.
Proportion of patients/teeth displaying furcation closure. | 12 months.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.
Proportion of patients/teeth displaying furcation closure. | 3 years.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.
Proportion of patients/teeth displaying furcation closure. | 5 years.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.
Proportion of patients/teeth displaying furcation closure. | 7 years.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.
Proportion of patients/teeth displaying furcation closure. | 10 years.
  Furcation closure defined as absence of clinically detectable furcation involvement degree >I.

SECONDARY OUTCOMES:
Changes in probing pocket depth. | 6 months.
  Reductions in PPD relative to baseline.
Changes in probing pocket depth. | 12 months.
  Reductions in PPD relative to baseline.
Changes in probing pocket depth. | 3 years.
  Reductions in PPD relative to baseline.
Changes in probing pocket depth. | 5 years.
  Reductions in PPD relative to baseline.
Changes in probing pocket depth. | 7 years.
  Reductions in PPD relative to baseline.
Changes in probing pocket depth. | 10 years.
  Reductions in PPD relative to baseline.
Changes in bleeding on probing. | 6 months.
  Reductions in BOP relative to baseline.
Changes in bleeding on probing. | 12 months.
  Reductions in BOP relative to baseline.
Changes in bleeding on probing. | 3 years.
  Reductions in BOP relative to baseline.
Changes in bleeding on probing. | 5 years.
  Reductions in BOP relative to baseline.
Changes in bleeding on probing. | 7 years.
  Reductions in BOP relative to baseline.
Changes in bleeding on probing. | 10 years.
  Reductions in BOP relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 6 months.
  Changes in clinical attachment levels relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 12 months.
  Changes in clinical attachment levels relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 3 years.
  Changes in clinical attachment levels relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 5 years.
  Changes in clinical attachment levels relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 7 years.
  Changes in clinical attachment levels relative to baseline.
Changes in vertical and horizontal clinical attachment level. | 10 years.
  Changes in clinical attachment levels relative to baseline.
Changes in marginal soft tissue levels. | 6 months.
  Changes in marginal soft tissue levels relative to baseline.
Changes in marginal soft tissue levels. | 12 months.
  Changes in marginal soft tissue levels relative to baseline.
Changes in marginal soft tissue levels. | 3 years.
  Changes in marginal soft tissue levels relative to baseline.
Changes in marginal soft tissue levels. | 5 years.
  Changes in marginal soft tissue levels relative to baseline.
Changes in marginal soft tissue levels. | 7 years.
  Changes in marginal soft tissue levels relative to baseline.
Changes in marginal soft tissue levels. | 10 years.
  Changes in marginal soft tissue levels relative to baseline.
Changes in radiographic bone levels. | 12 months.
  Changes in radiographic bone levels relative to baseline.
Changes in radiographic bone levels. | 3 years.
  Changes in radiographic bone levels relative to baseline.
Changes in radiographic bone levels. | 5 years.
  Changes in radiographic bone levels relative to baseline.
Changes in radiographic bone levels. | 10 years.
  Changes in radiographic bone levels relative to baseline.
Patient satisfaction assessed by visual analogue scale. | 6 months.
  Patient satisfaction as assessed on a 100 mm VAS.
Patient satisfaction assessed by visual analogue scale. | 12 months.
  Patient satisfaction as assessed on a 100 mm VAS.
Patient discomfort as expressed on a visual analogue scale. | 2 weeks.
  Patient discomfort following surgical therapy as expressed on a 100 mm VAS.
Patient discomfort as expressed on a visual analogue scale. | 6 months.
  Patient discomfort following surgical therapy as expressed on a 100 mm VAS.
Esthetic appreciation as expressed on a visual analogue scale. | 6 months.
  Esthetic appreciation as expressed on a 100 mm VAS.
Esthetic appreciation as expressed on a visual analogue scale. | 12 months.
  Esthetic appreciation as expressed on a 100 mm VAS.
Rate of adverse events. | 2 weeks.
  Impaired healing following surgical intervention.
Rate of adverse events. | 12 months.
  Impaired healing following surgical intervention.
Tooth loss. | 12 months.
  Event of tooth loss during follow-up.
Tooth loss. | 3 years.
  Event of tooth loss during follow-up.
Tooth loss. | 5 years.
  Event of tooth loss during follow-up.
Tooth loss. | 7 years.
  Event of tooth loss during follow-up.
Tooth loss. | 10 years.
  Event of tooth loss during follow-up.
Need for retreatment. | 12 months.
  Need for surgical retreatment of included site.
Need for retreatment. | 3 years.
  Need for surgical retreatment of included site.
Need for retreatment. | 5 years.
  Need for surgical retreatment of included site.
Need for retreatment. | 7 years.
  Need for surgical retreatment of included site.
Need for retreatment. | 10 years.
  Need for surgical retreatment of included site.
Change of inflammatory markers. | 2 weeks.
  Change of inflammatory markers measured in gingival crevicular fluid.
Change of inflammatory markers. | 6 weeks.
  Change of inflammatory markers measured in gingival crevicular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Karlsson, PhD, Study Director — Göteborg University
Locations (1):
- Department of Periodontology, Institute of Odontology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No